CLINICAL TRIAL: NCT04968795
Title: Effect of Heartfulness Corporate Wellness Program on Burnout Inventory Measurements
Brief Title: Heartfulness Meditation and Corporate Burnout
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Resolution Blue Labs Inc (Industry)
Collaborators: Heartfulness Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RBL-X Wellness_01
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Burnout; Meditation; Stress; Heartfulness
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Participate in filling the questionnaire but NOT the meditation/wellness session (control).
- Wellness Group: Participate in filling the questionnaire and the meditation/wellness session
  Interventions: Other: Heartfulness Meditation

INTERVENTIONS:
Other: Heartfulness Meditation — A four-week Heartfulness Wellness seminar, where people are exposed to Heartfulness Meditation and its meditation tools. Participants experience: Heartfulness Guided Relaxation, Heartfulness Meditation and Heartfulness Unwinding/Rejuvenation Technique.
  Groups: Wellness Group

SUMMARY:
The purpose of this study is to evaluate the effect of a 4-week heart-based meditation practice wellness workshop on burnout and emotional wellness in corporate employees. Corporate employees can be defined as individuals who work in large institutions with greater than 300 employees.

The specific aim of this study is to assess changes in scores measuring symptoms of emotional exhaustion, depersonalization, and personal accomplishment using the Maslach Burnout Index. We hypothesize that the meditation wellness practice will be associated with reduction in burnout for those who take part in the meditation program in comparison to the participants who did not meditate and participate in the wellness program.

ELIGIBILITY:
Inclusion Criteria:

* Adults above 18 years of age willing to participate in the study.

Exclusion Criteria:

* Individuals less than 18 years of age, active suicidal ideation, current or past diagnoses of serious psychotic disorders- schizophrenia, personality disorders and post-traumatic stress disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is reflective of the general population, who work in large corporations and have self-identified as having moderate to high levels of stress.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Differences in Burnout Scores | Week 0 & Week 4
  Assess the difference in burnout scores between both groups at week 0 and week 4.

SECONDARY OUTCOMES:
Changes in in scores measuring symptoms of emotional exhaustion, depersonalization, and personal accomplishment, using the Maslach Burnout Inventory. | Week 0 & Week 4
  Assess the difference in specific symptoms scores between both groups at week 0 and week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Kumar, MD/PhD Candidate, Principal Investigator — Resolution Blue Labs Inc; Aravindhan Ravindhran, MD, Principal Investigator — Resolution Blue Labs Inc; Arth Patel, MD Candidate, Principal Investigator — Resolution Blue Labs Inc
Locations (1):
- Resolution Blue Labs Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No